CLINICAL TRIAL: NCT06612177
Title: Latent Class Analysis and Phenotypes Identification of Surgical Site Infection in Elderly Patients After Non-cardiac Surgery---Based on a Prediction Model Established by Two Centers Large Sample
Brief Title: Elderly Patients Surgical Site Infection Phenotypes Identification
Status: Completed | Type: Observational
Sponsor: Weidong Mi (Other)
Responsible Party: Sponsor-Investigator, Weidong Mi, Depatment of Anesthesiology, The First Medical Center, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: PLAGH-AOC-L04
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Infection; Geriatrics; Prediction; Surgical Site Infection
Keywords: the elderly; prediction model; surgical site infection; latent class analysis
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study utilizes Latent Class Analysis (LCA) to identify phenotypes of Surgical Site Infection (SSI) in elderly patients following non-cardiac surgery. By analyzing data from two large cohorts, the research establishes a predictive model that uncovers independent risk factors for SSI, including age, hyperlipidemia, and surgical characteristics. The model, with AUCs ranging from 0.753 to 0.791 across cohorts, offers a calibrated prediction of SSI risk. Furthermore, LCA delineates four distinct SSI subphenotypes, highlighting a critical subgroup with a higher infection rate. This subgroup presents a complex interplay of risk factors, indicating the need for tailored preventive strategies. The study's findings contribute to a nuanced understanding of SSI in elderly surgical patients and pave the way for more targeted infection control measures.

DETAILED DESCRIPTION:
Backgrounds:

With the widespread use of prophylactic antibiotics during perioperative period and the continuous promotion of minimally invasive non-cardiac surgery type such as laparoscopic and thoracoscopic surgery, the incidence of superficial Surgical Site Infection (SSI) has been significantly reduced. Organ/deep SSI has become the dominant type of SSI. Currently, the classification of SSI is limited to the above location from shallow to deep, the epidemiological and clinical characteristics of SSI after non-cardiac surgery in elderly patients are still inadequately defined.

Objectives:

The investigators aimed to determine main risk factors for SSI after non-cardiac surgery among elderly patients in China and to further reveal the clinical attributes of those elderly patients afflicted with SSI.

Methods:

Potential risk factors for developing SSI were selected based on published data, clinical expertise, pathophysiological reasoning, and convenient considerations for future clinical applications. These SSI outcomes were rigorously calibrated by researchers complying with back-to-back principles following uniform diagnostic standards--European Perioperative Clinical Outcome (EPCO) definitions. According to the definitions, SSI in this study consists of three sites: superficial incision, deep incision, and organ/deep. The investigators define the occurrence of any of the above sites as SSI infection. Multivariable logistic regression analysis was used to identify risk factors for SSI. Data from population-based cohort of elderly patients undergoing non-cardiac and non-neurology surgery were used to derive the model. The risk prediction model was derived from the First Medical Center of the Chinese PLA General Hospital (January 2012 - August 2018). The investigators performed a nomogram, a complanation model based on the regression model with the graduated line segments as the main body. The discrimination was compared based on the AUC. The calibration was assessed by the calibration intercept and the slope. Decision curve analysis (DCA) was adopted to determine the nomogram's clinical usefulness and net benefit. Latent class analysis (LCA) was further used to explore the population features of SSI. LCA combines the latent variable theory with classified variables to explore the category latent variables behind statistically related classified explicit variables. Utilizing LCA, patients were classified into distinct cluster classifications, with each cluster's traits explained based on clinical factors. All continuous variables in the prediction model were treated as categorical variables before the LCA analysis. The number of categories was ascertained via the Bayesian information criterion (BIC). The lower BIC was also the elbow point which indicates better model fit. When determining the number of latent classes, clinical interpretations were taken into account. To demonstrate the combination of different risk factors in the prediction model, a chord chart and a characteristic data distribution map of subphenotypes were devised.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years;
2. Patients undergoing surgeries not involving local anesthesia.

Exclusion Criteria:

1. Patients undergoing neurosurgery or cardiac surgery;
2. Patients with preoperative infections (including pneumonia, SSIs, UTIs, and bloodstream infections);
3. Uncertain type of operation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The Training set included 42,532 elderly patients treated at the First Medical Center of the Chinese PLA General Hospital (PLAGH) from January 2012 to August 2018.
Sampling Method: Non-Probability Sample
Enrollment: 42532 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Elderly Patients Surgical Site Infection Phenotypes Identification | January 2012 - August 2018
  This study applies Latent Class Analysis to identify SSI phenotypes in elderly post-non-cardiac surgery patients, revealing four distinct subgroups with varying infection risks. The predictive model, validated across two cohorts, underscores the importance of tailored preventive strategies for high-risk subgroups, enhancing SSI management in elderly surgical patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital, Beijing, Beijing Municipality, China